CLINICAL TRIAL: NCT01363895
Title: Interventional Strategies in Treatment of Atrial Fibrillation: Percutaneous Closure of the Left Atrial Appendage Versus Catheter Ablation
Acronym: ISAR-AF
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Deutsches Herzzentrum Muenchen (Other)
Responsible Party: Isabel Deisenhofer, MD and Steffen Massberg, MD, Deutsches Herzzentrum München
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GER-EP-006
Record Dates: First submitted 2010-11-25; First posted 2011-06-02 (Estimated); Last update posted 2017-04-11 (Actual); Status verified 2017-04

CONDITIONS: Atrial Fibrillation
Keywords: atrial fibrillation; catheter ablation; percutaneous closure of LAA; intervention
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Percutaneous closure of LAA (Active Comparator): Percutaneous closure of LAA
  Interventions: Procedure: Percutaneous closure of LAA
- Catheter ablation of AF (Active Comparator): Catheter ablation of AF
  Interventions: Procedure: Catheter ablation of AF

INTERVENTIONS:
Procedure: Percutaneous closure of LAA — Percutaneous closure of LAA
  Arms: Percutaneous closure of LAA
Procedure: Catheter ablation of AF — Catheter ablation of AF
  Arms: Catheter ablation of AF

SUMMARY:
Atrial fibrillation (AF) is the most common sustained cardiac arrhythmia, associated with an increased risk of morbidity and mortality1. The management of AF patients is aimed at reducing symptoms and at preventing severe complications associated with AF. In the last years, two new strategies have emerged with different objectives. In the PROTECT AF study2, percutaneous closure of the Left Atrial Appendage (LAA) with a closure device provided an alternative strategy to oral anticoagulation for stroke prophylaxis. The AFFIRM trial3 has shown that drug-based management of AF with a rhythm-control strategy conferred no advantage over a rate-control strategy in cardiovascular mortality and might be associated with an increased noncardiovascular death rate4. Catheter ablation has gained a greater place in the rhythm control strategy, showing superiority in maintaining sinus rhythm in comparison with AAD5. However, in persistent AF, repeat ablation procedures are necessary in up to 70% of patients to achieve sinus rhythm at a long-term follow-up6-7.

This prospective, randomized trial will compare the percutaneous closure of the LAA combined with a rate-control strategy to catheter ablation in the management of patients with persistent AF. Patients who are eligible for catheter ablation as well as LAA closure device implantation and are willing to participate in the study will be randomly assigned to catheter ablation or percutaneous closure of the LAA by a closure device implantation in the relation 1:1. The primary endpoint of the study is a composite endpoint at 12 months of all cause death, thrombo-embolic events, major bleeding (BARC type 3), re-hospitalisation and severe symptoms due to arrhythmias. Secondary endpoints include a composite endpoint of bleeding, a composite endpoint of thrombo-embolic events, cardio-vascular mortality, total duration of hospitalisation, sustained discontinued anticoagulation, quality of life improvement, use of Antiarrhythmic Drugs (AAD), total costs, freedom from arrhythmia and average ventricular frequency in 7-day holter ECG at 12 months.

The objective of the study is to assess the superiority of percutaneous closure of the LAA combined with rate-control to catheter ablation in patients with oligosymptomatic AF.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with oligosymptomatic AF eligible for both interventions (CA and LAA closure device implantation).
2. Written, informed consent by the patient or her/his legally-authorized representative for participation in the study.
3. In women with childbearing potential a negative pregnancy test is mandatory.

Exclusion Criteria:

1. Left atrial thrombus
2. Other indication than AF for oral anticoagulation (valve prosthesis, pulmonary embolism, recurrent vein thrombosis)
3. Contraindication for oral anticoagulation
4. Severe valvular heart disease
5. Severe left ventricular systolic function (ejection fraction<30%)
6. Malignancies or other comorbid conditions (for example severe liver, renal and pancreatic disease) with life expectancy less than 12 months or that may result in protocol non-compliance.
7. Pregnancy (present, suspected or planned) or positive pregnancy test.
8. Patient's inability to fully cooperate with the study protocol.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2010-11; Primary Completion 2012-11 (Actual); Study Completion 2013-11 (Actual)

PRIMARY OUTCOMES:
A 12-month composite endpoint of all cause death, thrombo-embolic events, major bleeding BARC type III, re-hospitalisation and severe symptoms due to arrhythmias | 12 months

SECONDARY OUTCOMES:
The individual components of the primary endpoint | 12 months
Discontinuation of anticoagulation | 12 months
Quality of Life | 12 months
Use of Antiarrhythmic Drugs | 12 months
freedom from symptomatic arrhythmia | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Albert Schömig, MD, Study Chair — Deutsches Herzzentrum München; Steffen Massberg, MD, Principal Investigator — Deutsches Herzzentrum München; Isabel Deisenhofer, MD, Principal Investigator — Deutsches Herzzentrum München; Sonia Ammar, MD, Study Director — Deutsches Herzentrum München; Julia Goedel, MD, Study Director — Deutsches Herzzentrum München
Locations (1):
- Deutsches Herzzentrum München, Munich, Germany